CLINICAL TRIAL: NCT00137475
Title: A Phase I/II Feasibility/Efficacy Study Using Intensity-Modulated Radiation Therapy in Head and Neck (H&N) Cancer Patients to Permit Sparing of Parotid Gland Function
Brief Title: Using Intensity-Modulated Radiation Therapy to Permit Sparing of Parotid Gland Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA-15-0006 / 17086
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Head and Neck Cancer
Keywords: IMRT; head and neck cancer; parotid sparing
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Intensity-Modulated Radiation Therapy

SUMMARY:
Radiotherapy is the primary treatment modality or an important adjunct treatment for many patients with H&N carcinoma. Local control is directly related to dose and to the technical accuracy with which the dose is delivered to the target volume. Traditional radiotherapy techniques result in significant doses being delivered to normal tissues adjacent to the target, including the spinal cord and salivary glands. This leaves the patient with significant acute and late normal tissue toxicity that impacts on both the ability to tolerate the actual treatment and on the patient's long-term quality of life. Recently, the investigators have used static conformal multisegmental intensity modulated radiotherapy (IMRT) for a comprehensive irradiation of head and neck cancer with dose sparing of uninvolved tissues. This has resulted in substantial preservation of major salivary gland function in many patients with primary sites in the oral pharynx, oral cavity, nasopharynx, and pyriform sinus. While the investigators' results to date have shown promising preservation of salivary flow, they do not know whether patients treated with IMRT have similar local control rates as those treated with standard radiotherapy. Some investigators have raised the concern that by giving a low radiation dose to areas adjacent to the target volume there is a risk of undertreating the disease. On the other hand, the IMRT delivered with this protocol (called "simultaneous integrated boost", or SIB) may improve local control rates by delivering the same biologically effective dose in a shorter overall time period. This is a phase I/II trial which seeks to establish the efficacy of IMRT for H&N cancer treatment, and to further investigate the relationship between radiation dose to the parotid glands, salivary flow, and quality of life.

DETAILED DESCRIPTION:
Radiotherapy is the primary treatment modality or an important adjunct treatment for many patients with H&N carcinoma. Local control is directly related to dose and to the technical accuracy with which the dose is delivered to the target volume. Traditional radiotherapy techniques result in significant doses being delivered to normal tissues adjacent to the target, including the spinal cord and salivary glands. This leaves the patient with significant acute and late normal tissue toxicity that impacts on both ability to tolerate the actual treatment and on the patient's long-term quality of life. Recently, we have used static conformal multisegmental intensity modulated radiotherapy (IMRT) for comprehensive irradiation of head and neck cancer with dose sparing of uninvolved tissues. This has resulted in substantial preservation of major salivary gland function in many patients with primary sites in the oral pharynx, oral cavity, nasopharynx, and pyriform sinus. While our results to date have shown promising preservation of salivary flow, we do not know whether patients treated with IMRT have similar local control rates as those treated with standard radiotherapy. Some investigators have raised concern that by giving a low radiation dose to areas adjacent to the target volume there is a risk of undertreating disease. On the other hand, the IMRT delivered with this protocol (called "simultaneous integrated boost", or SIB) may improve local control rates by delivering the same biologically effective dose in a shorter overall time period (see below). This is a phase I/II trial which seeks to establish the efficacy of IMRT for H&N cancer treatment, and further investigate the relationship between radiation dose to the parotid glands, salivary flow, and quality of life. The specific objectives of the trial are as follows:

* To assess the local control rate and survival of patients treated with intensity-modulated radiotherapy using the simultaneous integrated boost (SIB) for regions at high risk of recurrence;
* To determine the patterns of failure of patients treated with IMRT+SIB;
* To assess the incidence of chronic grade 2 xerostomia after parotid-sparing IMRT using the RTOG grading scale;
* To assess quality of life of patients during and after IMRT using subjective xerostomia questionnaire and the University of Washington Quality of Life Head and Neck Symptom Questionnaire;
* To assess quantitative changes in salivary function before and after IMRT using sialometry (unstimulated and stimulated whole salivary flow rates).

Patients with squamous cell carcinoma of the H&N will be eligible provided they are over 18 years' age, AJCC stage I-IV with M0 and N0-2 disease, and KPS >=70%. Ineligibility criteria include previous cancer or H&N radiotherapy, salivary gland dysfunction, or unwilling to provide informed consent.

Methodology: All patients accrued to this study will have a series of pre-treatment evaluations, including history, physical, KPS evaluation, CT/MRI of the head and neck, chest x-ray or CT, dental examination, QOL assessment using the University of Washington QOL H&N symptom questionnaire (Hassan et al, 1993), and pre-treatment salivary flow measurements. All salivary flow measurements collected for this study will include unstimulated (resting) and stimulated (using citric acid solution), with a 5-minute collection time for each. Accrued patients will belong to one of two cohorts, which will determine the radiotherapy target volumes and dose levels: Group 1 - Patients who are treated with definitive radiotherapy (or chemoradiotherapy). The high dose region (PTV66) will consist of all areas of gross disease plus appropriate planning margin. The lower dose region (PTV54) will include PTV66 and all at-risk draining lymphatics of the neck. Group 2 - Patients treated with surgery and post-operative radiotherapy. The high-dose region (PTV60) will consist of the areas of previous gross disease and regions of the neck with metastatic lymph node involvement. The low-dose region (PTV54) will include PTV60 plus the remainder of the surgical bed and any additional regional lymphatic tissue considered to be at risk of harboring occult disease. All patients will be treated in 30 treatments (1 treatment per day, 5 days per week, for 6 weeks). PTV66 will receive 66 Gy, PTV54 will receive 54 Gy, etc. Thus different target regions will receive different doses per day (ranging from 1.8 to 2.2). In theory, giving high-risk regions a higher dose per day (hypofractionation) allows tumour cells less time to repopulate and should improve control rates (Fowler, 2000).

Investigations during and after treatment: Patients will have weekly toxicity assessments during radiotherapy. Follow-up after completion of RT will include history/physical, QOL assessment, and salivary flow collections. These assessments will be done at 4, 8, and 12 weeks, then every 1.5 months until 1 year. Follow-up beyond 1 year is at the physician's discretion but normally will involve visits every 3-4 months.

Statistical considerations: The sample size for this trial is based on the expected local control rate of similar patients treated with standard radiotherapy. For group 1 (patients treated with definitive radiotherapy) this is difficult to predict a priori because of the expected heterogeneity of stages and primary sites of accrued patients. However, stage I-II patients treated with RT alone, and selected stage III patients treated with chemoradiotherapy have 2-year local control rates of 70-80%. For group 2 (patients treated with surgery with high-risk features necessitating post-op RT), the expected local control rate is also approximately 70%. Assuming a power of 70%, significance of 5%, and a historical rate of local control of 75% (combined), the required number of patients to detect a 10% change in local control is 120.7. We will therefore accrue 120 patients, at an anticipated rate of 2-3 patients per month for 2-4 years.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell cancer of head and neck for radical/postoperative radiation therapy
* American Joint Committee on Cancer (AJCC) stage I-IV with M0 and N0-2 disease
* Karnofsky performance status (KPS) >= 70%

Exclusion Criteria:

* M1 or N3 disease
* Ineligibility for radiotherapy
* Recent malignancy
* Previous cancer or head and neck radiotherapy
* Salivary gland dysfunction
* Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2002-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
locoregional control rates
patterns of failure

SECONDARY OUTCOMES:
quality of life
saliva flow rates/xerostomia
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Rufus Scrimger, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada